CLINICAL TRIAL: NCT01855451
Title: TROG12.01 A Randomised Trial of Weekly Cetuximab and Radiation Versus Weekly Cisplatin and Radiation in Good Prognosis Locoregionally Advanced HPV-Associated Oropharyngeal Squamous Cell Carcinoma
Brief Title: Weekly Cetuximab/RT Versus Weekly Cisplatin/RT in HPV-Associated Oropharyngeal Squamous Cell Carcinoma
Acronym: HPVOropharynx
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROG 12.01; ACTRN12613000279729 (Registry Identifier: ANZCTR)
Record Dates: First submitted 2013-05-13; First posted 2013-05-16 (Estimated); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: HPV Positive Oropharyngeal Squamous Cell Carcinoma
Keywords: Human Papilloma Virus; HPV; Oropharyngeal; Squamous Cell; Carcinoma
MeSH Terms: conditions — Carcinoma | interventions — Cetuximab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiation Therapy + Cetuximab (Active Comparator): RT (70 Gy in 35 fractions, 5 days a week over 7 weeks) with weekly Cetuximab (400 mg/m2 loading dose IV prior to radiation, followed by weekly cetuximab 250 mg/m2 for the duration of the radiotherapy)
  Interventions: Drug: Cetuximab; Radiation: RT (70 Gy in 35 fractions)
- Radiation Therapy + Cisplatin (Active Comparator): RT(70 Gy in 35 fractions, 5 days a week over 7 weeks) with weekly Cisplatin (40 mg/m2 IV for the duration of the radiotherapy)
  Interventions: Radiation: RT (70 Gy in 35 fractions); Drug: Cisplatin

INTERVENTIONS:
Drug: Cetuximab
  Arms: Radiation Therapy + Cetuximab
Radiation: RT (70 Gy in 35 fractions)
Drug: Cisplatin
  Arms: Radiation Therapy + Cisplatin

SUMMARY:
A standard treatment for patients with head and neck cancer is radiation given with high doses of a chemotherapy drug called cisplatin, given every 3 weeks during the radiation. This treatment is effective but can significantly increase side effects such as difficulty with swallowing, a sore mouth, fatigue, hearing loss, ringing in the ears and kidney failure. In Australia, a commonly used treatment HPV-Associated Oropharyngeal Squamous Cell Carcinoma is a lower dose of cisplatin given weekly during the radiation. The high dose and low dose schedules result in a similar total dose of cisplatin being given during the radiation, but it is thought that the weekly schedule results in fewer side effects while maintaining effectiveness.

Another approach widely used around the world for patients with head and neck cancer, is to administer the antibody, cetuximab, weekly during radiation. Cetuximab has a very different side effect profile to cisplatin, and has been reported to result in less exacerbation of radiation related side effects. Both cetuximab and cisplatin can reduce the growth of a cancer and increase the effectiveness of radiation. Both cisplatin and cetuximab appear to be effective treatments in combination with radiation, but have not been directly compared.

The purpose of this study is to compare the treatment related side effects (both acute and longer term) between the cisplatin and cetuximab regimens. Both treatments would be given with the same dose of radiation therapy over 7 weeks. The results of this trial will help determine the optimal treatment for patients with HPV-Associated Oropharyngeal Squamous Cell Carcinoma.

DETAILED DESCRIPTION:
Human Papilloma Virus (HPV)-associated oropharyngeal squamous cell carcinoma (OPSCC) is increasing in incidence and has an improved prognosis compared to other head and neck malignancies when treated with standard combination chemoradiation.

The current standard regimen of high dose cisplatin and Radiation Therapy (RT) for head and neck cancer patients results in significant toxicity and is at the limits of tolerance. The excellent prognosis of patients with HPV-positive OPSCC raises concerns about overtreatment with the current standard of care, resulting in unnecessary acute and late morbidity.

Therefore, investigation of chemo-sparing or chemo-modified regimens with RT for HPV-associated OPSCC that do not compromise efficacy is warranted. A number of regimens less intensive than high dose cisplatin are being used in clinical practice for patients with good prognosis HPV OPSCC, but no comparative trials have been performed in this population. The trial population will be restricted to low risk HPV-associated OPSCC.

Trial Arms:

A- RT (70 Gy in 35 fractions, 5 days a week over 7 weeks) with weekly Cetuximab (400 mg/m2 loading dose IV prior to radiation, followed by weekly cetuximab 250 mg/m2 for the duration of the radiotherapy) B- RT(70 Gy in 35 fractions, 5 days a week over 7 weeks) with weekly Cisplatin (40 mg/m2 IV for the duration of the radiotherapy)

Hypothesis: In patients with locally advanced HPV-associated OPSCC, those treated with weekly cetuximab and conventionally fractionated radiotherapy will experience less acute symptom severity than patients receiving weekly cisplatin and conventionally fractionated radiotherapy.

Patients will be followed weekly during treatment, then at 1, 3, 5, 9, 13 weeks post-treatment and at months 6, 9, 12, 15, 18, 21, 24, 28, 32, 36, 42, 48, 54, and 60 post-completion of treatment. Follow-up for the trial will cease when the last patient accrued has a minimum of 2 years follow-up i.e. has attended the 24 months post-treatment review.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Has provided written Informed Consent for participation in this trial
3. Histologically confirmed squamous cell carcinoma of the oropharynx with p16 positive status confirmed locally by immunohistochemistry
4. Stage III (excluding T1-2N1) or stage IV (excluding T4, N3, and distant metastasis) if smoking history of < /=10 pack years. If > 10 pack years nodal disease must be N0 - N2a.
5. If an excisional biopsy has been performed, patients remain eligible for the study provided there is clinically measurable disease prior to commencing RT. The residual disease should still meet the stage criteria required for the trial e.g. excisional biopsy of a node with residual T3 primary, or tonsillectomy for T1 primary with residual > N2a nodes.
6. No prior treatment for oropharyngeal cancer
7. Adequate haematological, renal, and hepatic function as defined by,

   1. Absolute neutrophil count (ANC, segs + bands) > /= 1.5 x 109/L
   2. Platelet count > /= 100 x 109/L
   3. Total bilirubin < /= 1.5 x upper normal limit
   4. ALT < /= 2.5 x upper normal limit
   5. Calculated creatinine clearance (Cockcroft-Gault formula) or isotopic GFR > 55ml/min
8. ECOG performance status score of 0-1
9. Participants capable of childbearing are using adequate contraception and intend to continue use of contraception for at least 6 months following completion of treatment
10. Negative pregnancy test within 72 hours prior to randomisation of women who are of childbearing potential
11. Suitable for follow-up for at least 24 months as per trial protocol.
12. Sufficient proficiency in English, cognitive capacity and willingness to complete questionnaires

Exclusion Criteria:

1. History of unknown primary of the head and neck
2. T4, N3 or distant metastases
3. Smoking history >10 pack years with N2b or c nodal status
4. Women who are pregnant or lactating.
5. Previous radiotherapy to the area to be treated (excluding superficial radiotherapy for a cutaneous malignancy)
6. Previous cisplatin or carboplatin chemotherapy
7. Prior EGFR targeted therapy of any kind
8. Primary surgery to the affected area (excisional biopsy allowed)
9. Peripheral neuropathy > /= grade 2 (CTCAE v4.0)
10. Sensori-neural hearing impairment >= grade 2 (CTCAE v4.0, hearing impaired, not enrolled on a monitoring program) which may be exacerbated by cisplatin (Audiometric abnormalities without corresponding clinical deafness will not be grounds for exclusion)
11. Tinnitus > /= grade 2 (CTCAE v4.0)
12. History of interstitial lung disease or evidence of interstitial lung disease on pre-registration CT
13. History of myocardial infarction within 12 months prior to study entry, uncontrolled congestive heart failure, unstable angina, active cardiomyopathy, unstable arrhythmia, uncontrolled psychotic disorders, active serious infections, active peptic ulcer disease, immunosuppression due to post-organ transplantation or use of immunosuppressants for autoimmune disorders
14. Patients known to be HIV positive
15. Other cancer that was diagnosed:

    1. more than 5 years prior to current diagnosis with (i) subsequent evidence of disease recurrence or (ii) clinical expectation of recurrence is greater than 10% or
    2. within 5 years of the current diagnosis, with the exception of successfully treated basal cell or squamous cell skin carcinoma, in situ melanoma, or carcinoma in situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2013-06-03 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2023-08-23 (Estimated)

PRIMARY OUTCOMES:
Symptom Severity | 20 weeks
  The area under curve of symptom severity between weekly cisplatin and Radiotherapy Therapy (RT) versus weekly cetuximab and RT from baseline to week 20 (13 weeks post-completion of radiotherapy) as measured by M.D. Anderson Symptom Inventory - Head and Neck Module (MDASI-HN).

SECONDARY OUTCOMES:
Symptom severity | 24 months
  Symptom severity measured by MDASI-HN (Symptom Interference Score, Symptom Score, Symptom Clusters and individual item scores at individual time points)and by Functional Assessment of Cancer Therapy - Head and Neck (FACT-HN).
Interference of symptoms with daily life | 24 mths
  To compare interference of symptoms with daily life using the MDASI-HN Symptom Interference Score and Quality adjusted life years (QALYs) using the EQ-5D-5L
Psychological distress | 36 months
  To compare psychological distress measured by FACT-HN domain scores and depression and anxiety scales of Hospital Anxiety and Depression Scale (HADS)
Impact on Health Related Quality of Life | 36 months
Swallowing dysfunction | 12 months
  To compare swallowing dysfunction by Functional swallowing outcome (video fluoroscopy), CTCAE (v4.0) dysphagia, MDASI and FACT questionnaires, enteral feeding rates.
Speech and dietary function | 36 months
  To compare speech and dietary function as measured by the Performance Status Scale for Head & Neck Cancer Patients (PSS-HN)
Clinician-assessed acute and late toxicity | 60 months
  To compare clinician-assessed acute and late toxicity using toxicity grading (CTCAE v4.0) - reported as worst toxicity and as overall acute toxicity burden (T-score)
Rate of enteral feeding | 12 months
  To compare rate of enteral feeding at 12 months following treatment using Barnard's exact test for the comparison of two proportions
Hearing impairment | 24 months
  To compare hearing impairment, as measured by total score of the Hearing Handicap Inventory for adults, screening version (HHIA-S) and audiometry (results will be evaluated according to CTCAE 3 and 4 criteria, Brock criteria, Chang criteria and SIOP Boston Ototoxicity Scale).
Time to locoregional failure | 36 months
  To compare time to locoregional failure primarily determined by evidence of progression or recurrence clinically or radiologically
Failure-free survival | 36 months
  To compare failure-free survival by clinical and radioloigical assessments
Overall survival | 60 months
  To compare overall survival by clinical assessment.
Pattern of disease failure | 36 months
  Pattern of disease failure (locoregional [recurrence at primary tumour site and/or regional nodes], distant, both) as assessed radiologically.
Complete response rate | 20 weeks
  To compare FDG-PET-CT complete response rate at week 20
Cost of health resource utilisation | 24 months
  To compare cost of health resource utilisation via questionnaires EQ-5D-5L and RTOG return to work questionnaire.
Work status and time to return to work | 24 months
  To compare work status and time to return to work by RTOG questionnaire
Potential prognostic markers | 60 months
  To correlate several potential prognostic markers (including but not limited to EGFR protein level, EGFR copy number, ERCC1, plasma hepatocyte growth factor level, and plasma IL-8) with failure-free survival, overall survival and time to locoregional failure.

CONTACTS AND LOCATIONS:
Overall Officials: D Rischin, Dr, Study Chair — TROG and Peter MacCallum Cancer Centre
Locations (16):
- Australia (14):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - St George Hospital, Saint George, New South Wales
  - Riverina Cancer Care Centre, Wagga Wagga, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Womens Hospital, Herston, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Austin Hospital, Melbourne N., Victoria
  - Sir Charles Gairdner, Nedlands, Western Australia
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Palmerston North Hospital, Palmerston

REFERENCES:
- [Derived] Rischin D, King M, Kenny L, Porceddu S, Wratten C, Macann A, Jackson JE, Bressel M, Herschtal A, Fisher R, Fua T, Lin C, Liu C, Hughes BGM, McGrath M, McDowell L, Corry J. Randomized Trial of Radiation Therapy With Weekly Cisplatin or Cetuximab in Low-Risk HPV-Associated Oropharyngeal Cancer (TROG 12.01) - A Trans-Tasman Radiation Oncology Group Study. Int J Radiat Oncol Biol Phys. 2021 Nov 15;111(4):876-886. doi: 10.1016/j.ijrobp.2021.04.015. Epub 2021 Jun 4. PMID 34098030